CLINICAL TRIAL: NCT04756219
Title: Beneficial and Harmful Effects of Reducing Public Suicide Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Nathalie Oexle, Jun.-Prof. Dr. Nathalie Oexle, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 352/20
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Public Suicide Stigma
Keywords: Suicide; Stigma; General public; Suicide prevention
MeSH Terms: conditions — Suicide; Social Stigma; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Contact Video (Experimental): Participants randomized to this group will watch a video of a person talking about his recovery after attempting suicide.
  Interventions: Other: Contact Video
- Contact Text (Experimental): Participants randomized to this group will read a personal story of a person who survived a suicide attempt.
  Interventions: Other: Contact Text
- Education Video (Experimental): Participants randomized to this group will watch a video of a psychiatrist presenting facts about suicide and suicide prevention.
  Interventions: Other: Education Video
- Education Text (Experimental): Participants randomized to this group will read a text containing facts about suicide and suicide prevention.
  Interventions: Other: Education Text
- Control Contact (Placebo Comparator): Participants randomized to this group will read a personal story of a person who survived a heart attack.
  Interventions: Other: Contact Video; Other: Contact Text
- Control Education (Placebo Comparator): Participants randomized to this group will read a text containing facts about heart-attacks and their prevention.
  Interventions: Other: Education Video; Other: Education Text

INTERVENTIONS:
Other: Contact Video — No additional information necessary.
  Arms: Contact Video; Control Contact
Other: Contact Text — No additional information necessary.
  Arms: Contact Text; Control Contact
Other: Education Video — No additional information necessary.
  Arms: Control Education; Education Video
Other: Education Text — No additional information necessary.
  Arms: Control Education; Education Text

SUMMARY:
There is growing evidence that negative attitudes towards persons affected by suicide (i.e. persons who experience suicidality, persons who lost a loved one to suicide), so called public suicide stigma, is harmful for suicide prevention, for example by reducing social support, inhibiting help-seeking for suicidality and increasing distress as well as suicidality among stigmatized persons. Reducing public suicide stigma could therefore be an important factor of successful suicide prevention. However, reducing public suicide stigma could also be harmful, for example by increasing attitudes that suicidal behaviour is a normal and acceptable solution for crisis situations, which could decrease help-seeking for suicidality and encourage suicidal behaviour. This project will (1) develop four interventions (contact-based vs. education based, video vs. text) hypothesized to reduce public suicide stigma, (2) determine the efficacy of the four interventions with regard to reducing public suicide stigma, (3) identify additional harmful (e.g. normalization of suicidal behaviour) and beneficial intervention effects (e.g. improved attitudes to seek help) and (4) investigate pathways explaining intervention effects.

ELIGIBILITY:
Inclusion Criteria:

Participants need to be at least 18 years old, speak German and provide online informed consent.

Exclusion Criteria:

Persons who self-report to have experienced suicidality within three months before baseline will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Stigma subscale of the Stigma of Suicide Scale short form (SOSS-SF) | Immediately after the intervention (t1)
  Batterham al. (2013) The Stigma of Suicide Scale. Psychometric properties and correlates of the stigma of suicide. Crisis 34(1):13-21

SECONDARY OUTCOMES:
Stigma subscale of the Stigma of Suicide Scale short form (SOSS-SF) | Two weeks after the intervention (t2)
  Batterham al. (2013) The Stigma of Suicide Scale. Psychometric properties and correlates of the stigma of suicide. Crisis 34(1):13-21
Literacy of Suicide Scale (LOSS) | Immediately after the intervention (t1); Two weeks after the intervention (t2)
  Batterham et al. (2013) Correlates of suicide stigma and suicide literacy in the community. Suicide Life Threat Behav 43(4):406-417
Cognitions Concerning Suicide Scale (CCSS) | Immediately after the intervention (t1); Two weeks after the intervention (t2)
  Cwik et al. (2017) Measuring attitudes towards suicide: Preliminary evaluation of an attitude towards suicide scale. Compr Psychiatry 72:56-65
General help-seeking questionnaire suicidal ideation subscale (GHSQ-SI) | Immediately after the intervention (t1); Two weeks after the intervention (t2)
  Wilson et al. (2005) Measuring help-seeking intentions: Properties of the General Help-Seeking Questionnaire. Canadian Journal of Counselling 39(1):15-28
Current suicidality | Immediately after the intervention (t1); Two weeks after the intervention (t2)
  One item adapted from the PHQ-9 (Kroenke et al. 2001; "Do you currently experience thoughts that you would be better off dead or of hurting yourself?" response scale from 1 (not at all) to 7 (very much)
Positive and Negative Affect Schedule (PANAS), negative affect subscale | Immediately after the intervention (t1); Two weeks after the intervention (t2)
  Breyer & Bluemke (2016) Deutsche Version der Positive and Negative Affect Schedule PANAS (GESIS Panel). ZIS - GESIS Leibniz Institute for the Social Sciences
Patient Health Questionnaire (PHQ-2) | Two weeks after the intervention (t2)
  Löwe et al. (2005) Detecting and monitoring depression with a two-item questionnaire (PHQ-2). Journal of Psychosomatic Research 58(2):163-171

CONTACTS AND LOCATIONS:
Locations (1):
- Ulm University, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data available upon personal request.

REFERENCES:
- [Derived] Oexle N, Luhr M, Valacchi D, Rusch N. A web-based pilot randomized controlled trial to test the efficacy of education and contact-based interventions in reducing public suicide stigma. BMC Psychiatry. 2025 Jan 23;25(1):70. doi: 10.1186/s12888-024-06406-7. PMID 39849424